CLINICAL TRIAL: NCT04508829
Title: IMRT Combined With Concurrent Chemotherapy and Anti-EGFR Monoclonal Antibody in Locally Advanced Oropharyngeal Carcinoma Resistant to Induction Chemotherapy: a Multicenter Prospective Phase II Study.
Brief Title: Anti-EGFR Therapy With IMRT Concurrent Chemoradiotherapy in Locally Advanced OPC Resistant to Induction Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoshen Wang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPC-anti-EGFR-01
Record Dates: First submitted 2020-08-09; First posted 2020-08-11 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Oropharyngeal Carcinoma
Keywords: oropharyngeal carcinoma; IMRT; anti-EGFR monoclonal antibody; induced chemotherapy resistance
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-EGFR arm (Experimental): In the induction chemotherapy phase, TP regimen (Docetaxel 75mg/m2, D1 + DDP 25mg/m2, D1-3, repeat every 3 weeks) or TPF regimen (Docetaxel 75mg/m2, D1 + DDP 25mg/m2, D1-3+5-FU 750mg/m2, CIV, 120h, repeat every 3 weeks) will be used. Cetuximab 400mg/m2 will be used one week before radiotherapy and 250mg/m2/week during IMRT, or nimotuzumab 200mg/week; meanwhile, cisplatin 80mg/m2 will be used every 3 weeks.
  Interventions: Drug: Anti-EGFR monoclonal antibody

INTERVENTIONS:
Drug: Anti-EGFR monoclonal antibody — The patients will receive IMRT combined with anti-EGFR monoclonal antibody concurrent chemoradiotherapy in locally advanced oropharyngeal carcinoma with induced chemotherapy resistance. The specific treatment description is included in arm description.

SUMMARY:
This study is a prospective phase II trial which is designed to evaluate the efficacy and safety of IMRT combined with concurrent chemotherapy and anti-EGFR monoclonal antibody in locally advanced oropharyngeal carcinoma (OPC) with induced chemotherapy resistance.

Eligibility criteria include histologically confirmed locally advanced OPC according to the American Joint Committee on Cancer (AJCC) Staging System (the eighth edition); Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; at least one measurable lesion based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1; normal complete blood count, normal hepatic function and normal renal function. Prior induction chemotherapy with platinum was allowed.

Exclusion criteria include previous radiotherapy, a history of any other type of malignancy; pregnancy or lactation; allergy to anti-EGFR monoclonal antibody; obvious dysfunction of liver, renal, cardiac or lung function; uncontrolled infection; systemic metastasis or distant metastasis; patients with severe gastrointestinal diseases, and patients with mental disorders affecting patient participation in trial judgement.

The full-set pretreatment evaluation will be performed to every patient. All patients in this study will receive intensity-modulated radiation therapy (IMRT). The primary endpoints of this study is progression-free survival (PFS) and adverse events (AE) rate.

DETAILED DESCRIPTION:
This study is a prospective phase II trial which is designed to evaluate the efficacy and safety of IMRT combined with concurrent chemotherapy and anti-EGFR monoclonal antibody in locally advanced oropharyngeal carcinoma (OPC) with induced chemotherapy resistance.

Eligibility criteria include histologically confirmed locally advanced OPC with induced chemotherapy resistance according to the American Joint Committee on Cancer (AJCC) Staging System (the eighth edition); Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; at least one measurable lesion based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1; normal complete blood count (white blood cell counts ≥4×1012/L, hemoglobin level ≥100g/L and platelet counts ≥100×1012/L), normal hepatic function (total bilirubin level ≤1.5 mg/dl, alanine aminotransferase and aspartate aminotransferase levels ≤1.5 times the upper limit of normal) and normal renal function (creatinine ≤ 1.5 times the upper limit of normal). Prior induction chemotherapy with platinum was allowed.

Exclusion criteria include previous radiotherapy, a history of any other type of malignancy; pregnancy or lactation; allergy to anti-EGFR monoclonal antibody; obvious dysfunction of liver, renal, cardiac or lung function; uncontrolled infection; systemic metastasis or distant metastasis; patients with severe gastrointestinal diseases, and patients with mental disorders affecting patient participation in trial judgement.

The full-set pretreatment evaluation will be performed to every patient.All patients in this study will receive intensity-modulated radiation therapy (IMRT). In the induction chemotherapy phase, TP regimen (Docetaxel 75mg/m2, D1 + DDP 25mg/m2, D1-3, repeat every 3 weeks) or TPF regimen (Docetaxel 75mg/m2, D1 + DDP 25mg/m2, D1-3+5-FU 750mg/m2, CIV, 120h, repeat every 3 weeks) will be used. Cetuximab 400mg/m2 will be used one week before radiotherapy and 250mg/m2/week during IMRT, or nimotuzumab 200mg/week; meanwhile, cisplatin 80mg/m2 will be used every 3 weeks.

Adverse events (AEs) will be evaluated every week during CCRT based on the evaluation criteria of adverse reactions of CTCAE V4.0. Tumor response is assessed at the end of CCRT according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1. Radiation-related acute and late toxicities are graded according to the Radiation Therapy Oncology Group (RTOG). Late toxicities are evaluated beyond three months from the end of radiotherapy.

After the completion of CCRT, all patients will be followed up every 3 months during the first years, every 6 months for the following 2-5 years, and annually thereafter. Local recurrence is confirmed by oropharyngeal MRI or histological biopsy. Regional recurrence is confirmed by fine needle aspiration or surgical biopsy. Distant metastases is detected by imaging examinations including PETCT, bone Emission Computed Tomography (ECT), CT, MRI or confirmed by histological confirmation of biopsy.

The primary endpoints of this study is adverse events (AE) rate and progression-free survival (PFS). PFS is calculated from the date of enrollment to the date of disease progression or the date of death for any cause.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced OPC with Induced chemotherapy resistance;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Normal complete blood count;
* Normal hepatic function;
* Normal renal function (creatinine ≤ 1.5 times the upper limit of normal).

Exclusion Criteria:

* Previous radiotherapy;
* A history of any other type of malignancy;
* Pregnancy or lactation;
* Allergy to anti-EGFR monoclonal antibody;
* Obvious disfunction of liver, renal, cardiac or lung function;
* Un controlled infection;
* Systemic metastasis or distant metastasis;
* Patients with severe gastrointestinal diseases;
* Patients with mental disorders affecting patient participation in trial judgement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2016-01-01; Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 3-year PFS
  PFS is calculated from the date of the enrollment to the date of disease progression or the date of death for any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China